CLINICAL TRIAL: NCT03047538
Title: Fixed Combination for Lipid and Blood Pressure Control. Randomized Cross-over Study
Brief Title: Fixed Combination for Lipid and Blood Pressure Control
Acronym: FILIP
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient funds
Sponsor: Charles University, Czech Republic (Other)
Collaborators: University Hospital Olomouc (Other); University Hospital Pilsen (Other); General Teaching Hospital, Prague (Other); St. Anne (Unknown); Brno University Hospital (Other); Na Homolce Hospital (Other)
Responsible Party: Principal Investigator, Peter Wohlfahrt, Peter Wohlfahrt, MD, PhD, Charles University, Czech Republic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FILIP_V1.2
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Arterial Hypertension; Dyslipidemias; Blood Pressure; Lipid Metabolism Disorders
Keywords: Arterial hypertension; Dyslipidemia; Blood pressure control; Fixed combination
MeSH Terms: conditions — Hypertension; Dyslipidemias; Lipid Metabolism Disorders | interventions — Atorvastatin; Amlodipine; Perindopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Free combination (Active Comparator): Free combination of atorvastatin, perindopril and amlodipine will be given for 8 weeks. After 8 weeks free combination will be changed to fixed combination. The dose of each drug will be selected according to clinical judgement of each investigator, but can not be changed during the coarse of the study.
  Interventions: Drug: Atorvastatin, Amlodipine, Perindopril
- Fixed combination (Active Comparator): Fixed combination of atorvastatin, perindopril and amlodipine will be given for 8 weeks. After 8 weeks fixed combination will be changed to free combination. The dose of each drug will be selected according to clinical judgement of each investigator, but can not be changed during the coarse of the study.
  Interventions: Drug: Atorvastatin, Amlodipine, Perindopril

INTERVENTIONS:
Drug: Atorvastatin, Amlodipine, Perindopril — To compare free and fixed combination of atorvastatin, perindopril, amlodipine

SUMMARY:
The aim of this study is to compare the effect of fixed and free combination of atorvastatin/perindopril/amlodipine on blood pressure and lipid levels.

ELIGIBILITY:
Inclusion Criteria:

Patients with uncontrolled arterial hypertension (the average 24h blood pressure in the range 130/80 - 180/110 mmHg and / or daytime average blood pressure in the range 135/85-180/110 mmHg) and one of the following:

1. a very high cardiovascular risk and LDL-cholesterol> 1.8 mmol / l
2. a high cardiovascular risk and LDL-cholesterol> 2.5 mmol / l
3. Patient with a high or very high cardiovascular risk treated by lipidlowering therapy with statin

Exclusion Criteria:

1. hypersensitivity to perindopril or to other ACE inhibitors, amlodipine, atorvastatin, dihydropyridines or to or statins
2. angioneurotic edema in medical history (hereditary / idiopathic or associated with prior treatment with ACE inhibitors)
3. severe hypotension, shock, including cardiogenic shock
4. hemodynamically unstable heart failure
5. Active liver disease or unexplained persistent elevations of serum transaminases more than three times normal
6. Women of childbearing age without reliable contraception
7. pregnancy
8. breastfeeding
9. Patients with contraindications listed in the currently valid SP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood pressure control | 16 weeks - 8 weeks fixed and 8 weeks free combination atorvastatin, perindopril, amlodipine
  To compare the effect of fixed and free combination of atorvastatin/perindopril/amlodipine on 24h and in clinic blood pressure over the 16 weeks follow up.
Lipids control | 16 weeks - 8 weeks fixed and 8 weeks free combination atorvastatin, perindopril, amlodipine
  To compare the effect of fixed and free combination of atorvastatin/perindopril/amlodipine on LDL cholesterol levels over the 16 weeks follow up.

SECONDARY OUTCOMES:
Adherence | 16 weeks - 8 weeks fixed and 8 weeks free combination atorvastatin, perindopril, amlodipine
  1. To compare the effect of fixed and free combination of atorvastatin/perindopril/amlodipine on adherence evaluated by the Morisky medication adherence scale 8 and tablet counting over the 16 weeks follow up.
Blood pressure variability | 16 weeks - 8 weeks fixed and 8 weeks free combination atorvastatin, perindopril, amlodipine
  To compare the effect of fixed and free combination of atorvastatin/perindopril/amlodipine on 24h blood pressure variability over the 16 weeks follow up.
Arterial properties | 16 weeks - 8 weeks fixed and 8 weeks free combination atorvastatin, perindopril, amlodipine
  o compare the effect of fixed and free combination of atorvastatin/perindopril/amlodipine on arterial properties and central hemodynamic parameters measured during the 24 monitoring by the Mobilograph device over the 16 weeks follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Cardiovascular Prevention, Charles University Medical Faculty and Thomayer Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lawes CM, Vander Hoorn S, Rodgers A; International Society of Hypertension. Global burden of blood-pressure-related disease, 2001. Lancet. 2008 May 3;371(9623):1513-8. doi: 10.1016/S0140-6736(08)60655-8. PMID 18456100
- [Background] Stamler J, Wentworth D, Neaton JD. Prevalence and prognostic significance of hypercholesterolemia in men with hypertension. Prospective data on the primary screenees of the Multiple Risk Factor Intervention Trial. Am J Med. 1986 Feb 14;80(2A):33-9. doi: 10.1016/0002-9343(86)90158-0. PMID 3946459
- [Background] Gupta AK, Arshad S, Poulter NR. Compliance, safety, and effectiveness of fixed-dose combinations of antihypertensive agents: a meta-analysis. Hypertension. 2010 Feb;55(2):399-407. doi: 10.1161/HYPERTENSIONAHA.109.139816. Epub 2009 Dec 21. PMID 20026768
- [Background] Grimm R, Malik M, Yunis C, Sutradhar S, Kursun A; TOGETHER Investigators. Simultaneous treatment to attain blood pressure and lipid goals and reduced CV risk burden using amlodipine/atorvastatin single-pill therapy in treated hypertensive participants in a randomized controlled trial. Vasc Health Risk Manag. 2010 May 6;6:261-71. doi: 10.2147/vhrm.s7710. PMID 20479948
- [Background] Malekzadeh F, Marshall T, Pourshams A, Gharravi M, Aslani A, Nateghi A, Rastegarpanah M, Khoshnia M, Semnani S, Salahi R, Thomas GN, Larijani B, Cheng KK, Malekzadeh R. A pilot double-blind randomised placebo-controlled trial of the effects of fixed-dose combination therapy ('polypill') on cardiovascular risk factors. Int J Clin Pract. 2010 Aug;64(9):1220-7. doi: 10.1111/j.1742-1241.2010.02412.x. PMID 20653798
- [Background] Neutel JM, Bestermann WH, Dyess EM, Graff A, Kursun A, Sutradhar S, Yunis C. The use of a single-pill calcium channel blocker/statin combination in the management of hypertension and dyslipidemia: a randomized, placebo-controlled, multicenter study. J Clin Hypertens (Greenwich). 2009 Jan;11(1):22-30. doi: 10.1111/j.1751-7176.2008.00058.x. PMID 19125855
- [Background] PILL Collaborative Group; Rodgers A, Patel A, Berwanger O, Bots M, Grimm R, Grobbee DE, Jackson R, Neal B, Neaton J, Poulter N, Rafter N, Raju PK, Reddy S, Thom S, Vander Hoorn S, Webster R. An international randomised placebo-controlled trial of a four-component combination pill ("polypill") in people with raised cardiovascular risk. PLoS One. 2011;6(5):e19857. doi: 10.1371/journal.pone.0019857. Epub 2011 May 25. PMID 21647425
- [Background] Wald DS, Morris JK, Wald NJ. Randomized Polypill crossover trial in people aged 50 and over. PLoS One. 2012;7(7):e41297. doi: 10.1371/journal.pone.0041297. Epub 2012 Jul 18. PMID 22815989
- [Background] Indian Polycap Study (TIPS); Yusuf S, Pais P, Afzal R, Xavier D, Teo K, Eikelboom J, Sigamani A, Mohan V, Gupta R, Thomas N. Effects of a polypill (Polycap) on risk factors in middle-aged individuals without cardiovascular disease (TIPS): a phase II, double-blind, randomised trial. Lancet. 2009 Apr 18;373(9672):1341-51. doi: 10.1016/S0140-6736(09)60611-5. Epub 2009 Mar 30. PMID 19339045
- [Background] Thom S, Poulter N, Field J, Patel A, Prabhakaran D, Stanton A, Grobbee DE, Bots ML, Reddy KS, Cidambi R, Bompoint S, Billot L, Rodgers A; UMPIRE Collaborative Group. Effects of a fixed-dose combination strategy on adherence and risk factors in patients with or at high risk of CVD: the UMPIRE randomized clinical trial. JAMA. 2013 Sep 4;310(9):918-29. doi: 10.1001/jama.2013.277064. PMID 24002278
- [Background] Soliman EZ, Mendis S, Dissanayake WP, Somasundaram NP, Gunaratne PS, Jayasingne IK, Furberg CD. A Polypill for primary prevention of cardiovascular disease: a feasibility study of the World Health Organization. Trials. 2011 Jan 5;12:3. doi: 10.1186/1745-6215-12-3. PMID 21205325
- [Background] Cho EJ, Kim JH, Sutradhar S, Yunis C, Westergaard M; CRUCIAL trial investigators. Reduction in cardiovascular risk using a proactive multifactorial intervention is consistent among patients residing in Pacific Asian and non-Pacific Asian regions: a CRUCIAL trial subanalysis. Vasc Health Risk Manag. 2014 Mar 26;10:145-56. doi: 10.2147/VHRM.S54586. eCollection 2014. PMID 24707184